CLINICAL TRIAL: NCT01652456
Title: Alcohol and TObacco Consumption in Patients With Head and Neck Cancer : Interest of an Addiction Support
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ALTAKRA - 1205
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2014-08

CONDITIONS: Head and Neck Cancer; Lung Cancer
Keywords: addiction support; addiction specialist; lung cancer; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: Addiction support
- Group B (No Intervention)

INTERVENTIONS:
Other: Addiction support — one consultation with an addiction specialist
  Arms: Group A

SUMMARY:
This is a multicenter, interventional, randomized study for preventive and therapeutic strategies for patients with head and neck or Lung cancer; contribution of an addiction support

ELIGIBILITY:
Inclusion Criteria:

* first head and neck or lung cancer
* first support
* 18 ≤ age ≤ 60
* lives in Lille Metropolis
* having an addiction to alcohol and tobacco
* covered by health insurance
* signed informed consent

Exclusion Criteria:

* prior cancer
* mesothelioma and oesophageal cancer
* unable to undergo trail medical follow up (geographical, social and psychological reasons)
* pregnant or nursing woman
* patient under guardianship

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
systematic addiction consultation | 12 months after diagnosis
  difference between abstinence in group A and abstinence in group B

SECONDARY OUTCOMES:
progression free survival | 24 months after diagnosis
  median time between date of inclusion and date of first progression
overall survival | 24 months after survival
  median time between date of inclusion and date of death
alcohol and tobacco consumption | baseline, 3 months, 6 months and 12 months after diagnosis
  frequency of tobacco and alcohol consumption questionnaire : Fagerström, Alcohol Use Disorders Identification Test (AUDIT), Cut Down Annoyed Guilty Eye-Opener (CAGE-DETA), Cannabis abuse screening test (CAST), M.I.N.I.
alcohol + tobacco withdrawal and addiction support | 12 months after diagnosis
  difference between abstinence of group A and abstinence group B
addiction follow up | 24 months after diagnosis
  percentage of patient with a first addiction consultation, and willing to have a long term follow up

CONTACTS AND LOCATIONS:
Overall Officials: Corinne VANNIMENUS, MD, Study Director — Centre Hospitalier Régional et Universitaire
Locations (3):
- France (3):
  - Oscar Lambret Center, Lille
  - Centre Hospitalier Régional et Universitaire - Hopital CALMETTE, Lille
  - Centre Hospitalier Régional et Universitaire - Hopital HURIEZ, Lille